CLINICAL TRIAL: NCT00247195
Title: Culturally Congruent Care for Hispanic Outpatients With Major Depressive Disorder (MDD)
Brief Title: Effectiveness of Culturally Based Congruent Care in Treating Hispanics With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #4985; R34MH073087 (NIH); DSIR 82-SESC
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Depression
Keywords: Major Depression; MDD; Hispanic; Primary Care; Cultural Congruence
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culturally congruent assessment and treatment (Experimental): Outreach by phone to primary care patients interested in mental health referral. Engagement and evaluation approach conducted using the DSM-IV cultural formulation model. Same treatment choices as in control arm (medication, interpersonal psychotherapy, and combination treatment).
  Interventions: Behavioral: Culturally Congruent Assessment and Treatment
- Usual referral and treatment (Active Comparator): Usual referral procedure from primary care: PC clinician gives patient information on how to access mental health care at research site. Usual engagement and evaluation approach without using cultural formulation model. Same treatment choices (medication, interpersonal psychotherapy, and combination treatment) as in experimental arm.
  Interventions: Behavioral: Culturally Congruent Assessment and Treatment

INTERVENTIONS:
Behavioral: Culturally Congruent Assessment and Treatment — Referral, engagement, and treatment is done following the cultural formulation model in DSM-IV in which patients' views and expectations about depression treatment are included in the assessment and treatment process.

SUMMARY:
This study will develop and evaluate the effectiveness of a culturally based program that aims to facilitate entry, retention, and successful treatment in specialized mental health services for Hispanics with major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a type of depression that is characterized by a combination of symptoms that can interfere with the ability to work, study, sleep, eat, and enjoy activities that were once pleasurable. Studies have shown that individuals of Hispanic descent underutilize specialized mental health care services (SMHS), despite their need for it. In addition, Hispanic individuals have been associated with lower rates of retention in specialized mental health treatment. In particular, dropout rates from medication therapy for the treatment of MDD within SMHS are two to three times higher in Hispanics than in non-Hispanic whites. This study will develop and evaluate the effectiveness of a culturally-based program that aims to facilitate entry, retention, and successful treatment in specialized mental health services for Hispanics with MDD.

This open-label study will consist of four phases. Participants will be recommended for inclusion in the study upon receiving a diagnosis of MDD based on a standard health questionnaire completed in their primary care physician's office. Phase 1 of the study will entail an initial evaluation of the culturally congruent program of care for Hispanics with MDD (CCP-MDD). Participants will be placed in one of two focus groups, each composed of 8 to 10 people. One group will include individuals referred by their primary care physician. The other group will include family members of Hispanics with MDD. Discussions will focus on participants' understandings of depression-like illness, their treatment expectations for these conditions, and their perceived barriers to SMHS utilization. Information gathered in the focus groups will be used to develop a second version of CCP-MDD. Phase 2 of the study will evaluate the revised version of CCP-MDD and will include additional treatments with antidepressant medication, weekly interpersonal psychotherapy, or a combination of the two. Following treatment, participants will take part in a focus group, which will involve participant feedback.

Based on the information obtained in the focus groups and from clinical observations, a third version of CCP-MDD will be developed. In Phase 3, two sets of primary care offices will participate. One set will be assigned to the intervention arm, and receive the third version of the CCP-MDD intervention. A second set will be assigned to the control arm and receive usual referral to mental health services at the research site. All participants will be offered the same choice of treatments: antidepressant medication, weekly interpersonal psychotherapy, or a combination of the two. Treatment in both arms will be of the same duration, 18 wks. Focus groups will be held following treatment in order to obtain information about individuals' satisfaction or dissatisfaction with their care. Based on these findings, as well as clinical observations, a fourth and final version of CCP-MDD will be developed in Phase 4. All treatments will last a total of 18 weeks. A follow-up session will be held at Week 30 to assess depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

PHASE 1 FOCUS GROUP 1:

* Self-identifies as Hispanic
* Screened positive for MDD during the previous study (WH-PCDP), but was unable to participate in that study due to ongoing depression treatment at the time
* Spanish-speaking

PHASE 1 FOCUS GROUP 2:

* Self-identifies as Hispanic
* Family member of a patient with MDD who participated in the previous study (WH-PCDP)
* Spanish-speaking

PHASES 1-3:

Pre-Engagement Phase

* Self-identifies as Hispanic
* Spanish-speaking
* Positive screen for MDD on the Patient Health Questionnaire (PHQ) and a preliminary diagnosis of MDD from the primary care physician during a standard medical interview

Treatment Phase

* Meets DSM-IV criteria for MDD
* Score of at least 16 on the Hamilton Depression Scale (HAM-D17) at the time of study entry
* Willing to abstain from any other type of specialized mental health services for the duration of the treatment (participants in general health care or participating in folk/spiritual healing practices are expected to continue these during the study)
* Ability to tolerate a drug-free period (2 weeks for most medications; 4 weeks for fluoxetine) if on an ineffective psychotropic medication; if current medication is effective, participants will not be asked to discontinue it (zolpidem for insomnia is also a permitted medication)
* Agrees to use an effective form of contraception for the duration of the study

Exclusion Criteria

PHASE 1 FOCUS GROUP 1:

* Comorbid medical or psychiatric conditions that may prevent focus group participation (e.g., substance use disorders, psychosis, unstable medical conditions)
* Active suicidal or homicidal ideation that may pose a danger to oneself or others

PHASE 1 FOCUS GROUP 2:

* Comorbid medical or psychiatric conditions that may prevent focus group participation (e.g., substance use disorders, psychosis, unstable medical conditions)

PHASES 1-3:

Pre-Engagement Phase

* Declines referral by a primary care physician to specialized mental health services
* Comorbid medical or psychiatric conditions that may prevent safe study participation (e.g., substance use disorders, psychosis, unstable medical conditions)
* Active suicidal or homicidal ideation that may pose a danger to oneself or others

Treatment Phase

* History of schizophrenia, bipolar disorder, schizoaffective disorder, depression with psychotic symptoms, or organic brain syndromes
* Clinically unstable medical disease, including glaucoma
* Blood pressure higher than 150/90
* Pregnant or breastfeeding
* Current or past history of seizure disorder (except febrile seizure in childhood)
* Meets DSM-IV criteria for alcohol or substance abuse or dependence (except nicotine) within the 6 months prior to screening
* Use of monoamine oxidase inhibitors (MAOIs) or fluoxetine within 4 weeks prior to screening, or use of other selective serotonin reuptake inhibitors (SSRIs), antidepressants, neuroleptics, mood stabilizers, buspirone, benzodiazepines, or other psychotropic drugs, except zolpidem for insomnia within 2 weeks prior to screening
* Currently receiving formal psychotherapy from a mental health provider, whether or not the focus of the therapy is MDD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2005-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Entry into specialty mental health care from primary care | Measured at study completion
Entry into treatment for major depressive disorder after evaluation | Measured at study completion
Dropout from stepped care | Measured throughout the study

SECONDARY OUTCOMES:
Score on the Hamilton Depression Scale (17-item) | Measured at Week 30
Score on the Clinical Global Impression Scale | Measured at Week 30
Score on the Working Alliance Inventory | Measured at Week 18
Score on the Client Satisfaction Questionnaire | Measured at Week 18
Score on the Side Effects Checklist | Measured at Week 18
Score on the Quality of Life Index | Measured at Week 30
Score on the Social Adjustment Scale - Self-report version | Measured at Week 30
Score on the Client Satisfaction Questionnaire | Measured at Week 30
Score on the Nervios Treatment Scale | Measured at Week 30
Score on the Working Alliance Inventory | Measured at Week 30
Score on the Clinical Global Impression Scale - Patient version | Measured at Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Lewis-Fernandez, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute - Hispanic Treatment Program, New York, New York, United States